CLINICAL TRIAL: NCT03756376
Title: The Relationship Between IRRIV and RFR Under Pathologic Conditions
Acronym: IRRIV-RFR
Status: Completed | Type: Observational
Sponsor: Ospedale San Bortolo di Vicenza (Other)
Responsible Party: Principal Investigator, Sara Samoni, Medical Doctor, Ospedale San Bortolo di Vicenza
Other Study IDs: 35/14
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IRRIV and RFR: Enrolled patients will receive IRRIV test and RFR assessment. RFR will be evaluated through a protein loading test. (1.2 g of protein/Kg of body weight) performed with cooked beef. The RFR was then defined as the difference between the highest CrCl obtained after the protein load and the baseline CrCl measured on rest conditions. Concerning the IRRIV test, a weight of 10% of the patient's body weight is applied on the abdominal wall. RRIs is recorded in a middle interlobular artery, every minute for 10 minutes during the echo-renal stress test. The lowest RRI reached is taken as reference (stress RRI). The IRRIV is defined as the percentage difference between baseline RRI and stress RRI

SUMMARY:
The assessment of renal functional reserve (RFR) has been proposed for the risk stratification of patients undergoing potentially nephrotoxic procedures. The present pilot study is designed to explore the correlation between IRRIV and RFR under pathologic conditions.

DETAILED DESCRIPTION:
Renal functional reserve (RFR) represents the capacity of the kidney to increase glomerular filtration rate (GFR) in response to certain physiological or pathological stimuli or conditions.

RFR is calculated as the difference between the measured maximum GFR achieved through a renal stress test and the baseline GFR measured in rest conditions. In clinical practice, the most common renal stress test is performed as a standardized protein loading test. Recently, in a pilot study, the investigators demonstrated a significant correlation between RFR and the intra-parenchymal renal resistive index variation (IRRIV) during an echo renal stress test in a cohort of healthy volunteers. IRRIV test has proven to be rapid, safe, bedside and easy to perform and it might represent a preliminary test in screening patients' RFR.The present pilot study is designed to explore the correlation between IRRIV and RFR under pathologic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Estimated GFR (CKD-EPI) greater than or equal to 60 mL/min/1.73 m2
* Scheduled cardiac surgery with cardiopulmonary bypass (coronary artery bypass, valve replacements, combined or other operations).

Exclusion Criteria:

* Age less than 18 years old
* Pregnancy
* Ultrasound evidence of morphological kidney abnormalities and/or renal artery stenosis
* Nonsteroidal anti-inflammatory drugs (NSAIDs)
* Contrast media in the 2 days before the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery with cardiopulmonary bypass (coronary artery bypass, valve replacements, combined or other operations)
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2016-01-13 (Actual)

PRIMARY OUTCOMES:
Correlation between IRRIV test and RFR in cardiac surgery patients | Change from baseline to 60 minutes
  IRRIV test and RFR will be determined and a relationship will be assessed

SECONDARY OUTCOMES:
Concordance between IRRIV test and RFR in cardiac surgery patients | Change from baseline to 60 minutes
  Concordance between presence of RFR (i.e. a RFR≥15ml/min/1.73m2) and a positive/uncertain/negative IRRIV is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, Study Director — Ospedale San Bortolo di Vicenza

REFERENCES:
- [Result] Samoni S, Nalesso F, Meola M, Villa G, De Cal M, De Rosa S, Petrucci I, Brendolan A, Rosner MH, Ronco C. Intra-Parenchymal Renal Resistive Index Variation (IRRIV) Describes Renal Functional Reserve (RFR): Pilot Study in Healthy Volunteers. Front Physiol. 2016 Jul 6;7:286. doi: 10.3389/fphys.2016.00286. eCollection 2016. PMID 27458386
- See also: SSamoni ppt — https://www.youtube.com/watch?v=9V4RoWvL9cs